CLINICAL TRIAL: NCT07246902
Title: MOVE - Mobilization and Outcomes After VEnous Closure - A Prospective Registry of Real-World Outcomes/Usage/Evidence for the MYNX CONTROL™ VENOUS Vascular Closure Device 6F-12F
Brief Title: Mobilization and Outcomes After Venous Closure
Acronym: MOVE
Status: Recruiting | Type: Observational
Sponsor: Cordis US Corp. (Industry)
Collaborators: NAMSA (Other)
Responsible Party: Sponsor
Other Study IDs: P25-8302
Record Dates: First submitted 2025-11-13; First posted 2025-11-24 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Venous Vascular Closure; Electrophysiology Study
Keywords: Electrophysiology Study; Venous closure; Venous access closure; Vascular access closure; Venous Vascular Closure; Vascular closure device; MYNX CONTROL VENOUS; MOVE Registry; MOVE; Cardiac Catheterization; MYNX

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- MCV VCD Treatment: Subjects who undergo catheter-based procedures utilizing 6F to 12F inner diameter procedural sheaths, with single or multiple venous access sites in one or both limbs, and have their venous access site(s) closed with MYNX CONTROL™ VENOUS VCD 6F-12F per IFU.
  Interventions: Device: MYNX CONTROLTM VENOUS Vascular Closure Device

INTERVENTIONS:
Device: MYNX CONTROLTM VENOUS Vascular Closure Device — The MYNX CONTROLTM VENOUS (MCV) Vascular Closure Device (VCD) 6F-12F is indicated for use to seal femoral venous access sites while reducing times to hemostasis and ambulation in patients who have undergone diagnostic or interventional endovascular procedures utilizing 6F to 12F procedural sheaths, with single or multiple access sites in one or both limbs.
  MCV VCD is designed to achieve femoral vein hemostasis via delivery of the GRIP TECHNOLOGY™ sealant (an extravascular, water-soluble synthetic hydrogel), using a balloon catheter in conjunction with a standard procedural sheath. The sealant is made of a polyethylene glycol (PEG) material which expands upon contact with subcutaneous fluids to seal the venotomy and is resorbed by the body within 30 days.
  The MCV VCD is supplied with a 10ml locking syringe used for balloon inflation and deflation. The catheter shaft has a silicone lubricant to facilitate insertion and withdrawal into compatible sheaths.

SUMMARY:
The primary objective of this post-market registry is to collect real-world outcomes and evaluate usage practice of MYNX CONTROL™ VENOUS (MCV) Vascular Closure Device (VCD) 6F-12F in sealing femoral venous access sites in patients who have undergone endovascular procedures in a real-world setting.

DETAILED DESCRIPTION:
The study is a single-arm, prospective, multi-center, observational, real-world registry of venous access site closures utilizing MYNX CONTROL™ VENOUS VCD 6F-12F following endovascular procedures. The study will enroll approximately 300 subjects in approximately 15 study sites in the United States.

ELIGIBILITY:
Inclusion Criteria

1. Able and willing to provide informed consent and to complete a follow-up visit at 14 ± 7 days post-procedure.
2. Individuals undergoing catheter-based procedures utilizing 6F to 12F inner diameter procedural sheaths, with single or multiple venous access sites in one or both limbs.
3. Individuals who are candidates to have their venous access site(s) closed with MYNX CONTROL™ VENOUS VCD 6F-12F per IFU.
4. At the time of enrollment, the Investigator deems the subject a candidate for same-day discharge (SDD) per standard of care (no procedure related events/complications e.g., no new pericardial effusion, post-procedure diuresis not needed, etc.).

Exclusion Criteria

1. Presence of bruit, palpable aneurysm, significant candida or groin infection.
2. Prior to closure, presence of hematoma in the accessed limb.
3. Currently involved in any other clinical trial that may interfere with the outcomes of this study as determined by the Investigator.
4. Planned use of other closure devices or techniques other than MYNX CONTROL™ VENOUS VCD 6F-12F.
5. Life expectancy <12 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study includes patients who undergo catheter-based procedures utilizing 6F to 12F inner diameter procedural sheaths, with single or multiple venous access sites in one or both limbs, and have their venous access site(s) closed with MYNX CONTROL™ VENOUS VCD 6F-12F per IFU.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with same day discharge (SDD) and without subsequent hospitalization/intervention for access-site complications | From time of index procedure through end of following day (within 48 hours)
  Rate of patients who successfully received a study device at all access sites and had SDD without subsequent hospitalization/intervention for access-site complications either same day post-discharge or the next day
Rate of access-site complications | From time of study device introduction at first access site through 14 days post-procedure
  Rate of access-site complications, assessed per standard of care, through 14 days post-procedure, including:
  * Access Site-Related Hematoma > 6 cm documented by ultrasound
  * Local Access Site Infection confirmed by culture and sensitivity, treated with intramuscular or oral antibiotics
  * Allergic Reaction
  * Access site-related bleeding requiring transfusion, surgical intervention, or rehospitalization
  * Pulmonary embolism requiring surgical or endovascular intervention and/or resulting in death, to be confirmed by CT pulmonary angiography, lung ventilation/perfusion scan (VQ scan), or autopsy
  * DVT requiring pharmaceutical or surgical intervention

OTHER OUTCOMES:
Time to Ambulation | From end of index procedure until time before hospital discharge (usually within ~24 hours of procedure)
  Defined as elapsed time (in hours) between removal of the final MCV VCD and when subject stands and walks 20 feet without evidence of rebleeding from any femoral venous access site.
Time to Discharge | From end of index procedure until time of hospital discharge (usually within ~24 hours of procedure)
  Defined as the elapsed time (in minutes) between removal of the final MCV VCD and when the subject is discharged from the hospital, as recorded on the discharge order.
Time to Hemostasis | From time of index procedure until time before hospital discharge (usually within ~24 hours of procedure)
  Defined as elapsed time (in minutes) between removal of each MCV VCD and first observed and confirmed venous hemostasis (per access site analysis).
SDD sustained MCV VCD success | From end of index procedure through 14 days post-procedure
  Defined as the proportion of subjects who did not require hospital intervention within 14 days post-procedure due to access site-related complications
Device success evaluated at the end of the procedure | End of index procedure
  Defined as the ability to deploy the delivery system and deliver the PEG component to achieve hemostasis at each access site
Procedural Success | From end of index procedure through 14 days post-procedure
  Defined as the attainment of final hemostasis at all venous access sites without major venous access site closure-related complications through 14 days
Procedural Time | Index procedure
  Defined as time of first sheath insertion until the time of removal of final MCV VCD.
Recovery room time | From time of transfer to recovery room post-discharge to time of discharge (usually within ~24 hours of procedure)
  Defined as elapsed time (in minutes) between when the subject is transferred to recovery and when the subject is discharged from the hospital, as recorded on the discharge order.
Analysis of Cost Effectiveness - Comprehensive summary of clinical outcomes, resource utilization, economic proxies, patients reported outcomes and CPT codes | From start time of index procedure through 14 days post-procedure
  An analysis of cost effectiveness will be performed based on a summary of key clinical outcomes, resource utilization, economic proxies, patients reported outcomes and CPT codes
Incidence of urinary catheter usage | From start time of index procedure through end time of index procedure
  Number/rate of patients with urinary catheters used during the procedure
Rate of protamine usage | From start time of index procedure through end time of index procedure
  Rate of protamine usage during the procedure
Medication Usage | From pre-procedure though study exit/follow-up visit (14 +/- 7 days post-procedure)
  Rate of patients who are administered anti-platelet, anti-coagulant, anti-thrombotic, local anesthetic, protamine or pain medication)

CONTACTS AND LOCATIONS:
Locations (1):
- KC Heart and Rhythm Institute, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided